CLINICAL TRIAL: NCT04902586
Title: The Clinical Effect and Safety of Radiotherapy Concurrent of TTFields in the Treatment of Post-operation Patients With Glioblastoma.
Brief Title: Effect of Radiotherapy Concurrent of TTFields in Patients With Glioblastoma
Acronym: ECTG001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZhongnanH ECTG001
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Glioma; Glioblastoma
Keywords: glioblastoma; TTFields; radiotherapy
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E group (Experimental): All patients received chemoradiotherapy (CRT) ( PTV-GTV: 60Gy at 2.0Gy per fraction, 5 fractions per week for 6 weeks; PTV-CTV: 54Gy at 1.8Gy per fraction, 5 fractions per week for 6 weeks) with a Temozolomide (TMZ) regimen（75mg/m2 per day during RT）and TTFields therapy during RT. The TTFields therapy started on the day the radiotherapy started.
  Interventions: Device: TTFields
- C group (No Intervention): All patients received chemoradiotherapy (CRT) ( PTV-GTV: 60Gy at 2.0Gy per fraction, 5 fractions per week for 6 weeks; PTV-CTV: 54Gy at 1.8Gy per fraction, 5 fractions per week for 6 weeks) with a Temozolomide (TMZ) regimen（75mg/m2 per day during RT）

INTERVENTIONS:
Device: TTFields — The TTFields, consisting of low-intensity, 200 kHz frequency, alternating electric fields, was delivered (≥ 18 hours/d) via 4 transducer arrays on the shaved scalp and connected to a portable device.
  Arms: E group

SUMMARY:
TTFields has been approved by the FDA for the treatment of patients with glioblastoma multiforme. However, the clinical effect and safety of radiotherapy concurrent of TTFields is not definite. In this study, the investigators conduct a phase II clinical trial to evaluate the efficacy and safety of this strategy.

DETAILED DESCRIPTION:
the investigators plan to recruit 30 patients to evaluate the efficacy and safety of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* performance status of 0-1 (Eastern Cooperative Oncology Group performance status)
* histologically confirmed glioblastoma
* no cerebrospinal fluid and distant metastatic disease.

Exclusion Criteria:

* with a history of brain radiotherapy
* severe hepatic and renal dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-19 (Estimated); Primary Completion 2021-12-19 (Estimated); Study Completion 2022-07-19 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 1 year
  the length of time after primary treatment for glioblastoma ends that the patient survives without any signs or symptoms of glioblastoma.

SECONDARY OUTCOMES:
Overall survival | 2 years
  The length of time from the date of diagnosis to death from cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jianyin Huang, MD, Study Chair — Wuhan University
Locations (1):
- Zhongnan hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No